CLINICAL TRIAL: NCT00244699
Title: A Mindfulness-Based Intervention for Youth With Concurrent Disorders
Brief Title: Integrating Mindfulness-Based Skills Training Into Brief Outpatient Treatment for Substance Abusing Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200/2005
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Substance Abuse; Drug Addiction
Keywords: youth; drug addiction; substance abuse; mindfulness; motivational interviewing; brief treatment; skills training; group therapy; emotion regulation
MeSH Terms: conditions — Substance-Related Disorders; Emotional Regulation

INTERVENTIONS:
Behavioral: MI Alone or Plus Mindfulness-Based Skills Training

SUMMARY:
The proposed study will evaluate the clinical effectiveness of integrating mindfulness-based skills training into a standardized brief group intervention for youth (ages 16 to 24) identified as having problematic substance use. Forty youth (N = 20 per group) will be randomized to one of two treatment conditions: 1) a standardized 4-week brief treatment for problematic substance use (treatment as usual; TAU) or 2) standardized brief treatment (TAU) augmented with a mindfulness skills training component based primarily on the mindfulness module described in Linehan's (1993b) Dialectical Behavior Therapy skills group training. It is expected that, compared to the TAU, the mindfulness-based group plus TAU will produce superior outcomes on the following primary outcome measures: number of substance use days, confidence to resist urges to use substances, and mindfulness skills. Secondary outcomes that will be examined include severity of consequences of use, general psychiatric symptoms, self-compassion, emotion dysregulation, and transfer to further treatment.

DETAILED DESCRIPTION:
For a wide range of clinical conditions (e.g., depression, anxiety, chronic pain, and stress-related health problems), the integration of mindfulness based interventions into clinical treatment has yielded positive benefits (e.g., Kabat-Zinn, 1990; Segal, Williams, & Teasdale, 2002; see Appendix II for a list of references for the study). Recently, researchers have found mindfulness skills training to have a number of beneficial treatment implications for substance abuse in adults (e.g., Alterman, A.I., Koppenhaver, J, Mulholland, E, Ladden, L, & Baime M. (2004); Breslin, Zack, & McMain, 2002; Marcus, 2005; Marlatt, 2005; Marlatt & Kristeller, 1999). Although researchers have recommended that mindfulness be implemented as an adjunctive treatment for addictions, including the early stages of substance use treatment (Breslin et al., 2002; Marcus, 2001; 2003; 2005), few studies have explored whether incorporating mindfulness skills training yields incremental benefits over standard treatments alone, or whether mindfulness skills have clinical utility during the early stages of substance abuse treatment. Moreover, no studies have explored the relative benefits of incorporating mindfulness skills training into the treatment of problematic substance use among transition-age youth, an age group at heightened risk for the development of addiction and mental health problems (Beitchman, Adlaf, Douglas, Atkinson, Young, et al., 2001). The integration of mindfulness into youth substance abuse treatment would be expected to yield beneficial effects given the developmental patterns of impulsivity and emotion dysregulation frequently characterizing this population (Winters, 1999). Researchers using the mindfulness paradigm have proposed that one of the key beneficial mechanisms produced by mindfulness is emotional regulation (e.g., Linehan, 1993a, 1993b; see Roemer, 2003). By increasing mindfulness, and thereby emotion regulation, therapy clients undergoing mindfulness skills training would be expected to experience an enhanced capacity to resist impulses to act on substance use urges (Breslin et al., 2002). Thus, when integrated into treatment as usual, mindfulness skills training would be expected to have positive, incremental effects on clients' abilities to reduce their level of substance use over the course of substance abuse treatment.

This study will address the question: Does the integration of mindfulness-based skills training into a standardized brief substance abuse treatment (TAU) for youth enhance treatment outcomes compared to standardized treatment (TAU) alone? Clinical outcomes will be compared for youth randomized to one of two treatment conditions: a) a TAU control condition, consisting of an evidence-based, standardized brief treatment group delivered in approximately 2-hour sessions once per week over four weeks (i.e., the First Contact group; Breslin, Li, Sdao-Jarvie, Tupker, & Ittig-Delan, 2002), and b) an experimental treatment condition, consisting of the TAU enhanced with a mindfulness skills training component based primarily on the mindfulness module described in Linehan's (1993) Skills Training Manual for Treating Borderline Personality Disorder (Linehan, 1993b), and recent adaptations of these skills for substance use problems (McMain, Dimeff, Sayrs, Davis, & Linehan, 2005), and youth populations (Miller, Rathus, Landsman, & Linehan, in press). This study will explore whether, when compared to the TAU, the treatment augmented with mindfulness skills training will have a beneficial impact on clinical outcomes, including the confidence to resist substance use urges, number of substance use days, and the development of mindfulness skills.

The primary hypotheses are that, compared to TAU, the group receiving treatment enhanced with mindfulness skills training will report the following: (1) a lower number of substance use days, (2) greater confidence to resist urges to use substances, (3) a higher level of mindfulness skills. Secondary analyses will explore the extent to which the experimental condition is related to beneficial effects on the following: (1) negative consequences of substance use, (2) psychiatric symptoms, (3) difficulties with emotion regulation, (4) self-compassion, (5) rates of transfer to further treatment, and (6) premature treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* One or more indicators of problematic substance use over the past 60 days and brief group treatment for problematic substance use is indicated

Exclusion Criteria:

* Current active or unmanaged psychosis, bipolar disorder, self-harm or suicidality

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2005-10; Study Completion 2007-04

PRIMARY OUTCOMES:
The following will be measured T1 (pre-treatment)to T4(3-month follow-up), as well as at each weekly tx session:
number substance use days
confidence to resist urges to use substances
mindfulness skills

SECONDARY OUTCOMES:
The following will be measured T1 (pre-treatment) to T4(3-month follow-up):
negative consequences of substance use
psychiatric symptoms
difficulties with emotion regulation
self-compassion
The following will be measured post-treatment or following drop-out from treatment:
rates of transfer to further treatment
reasons for premature treatment termination

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Vettese, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada